CLINICAL TRIAL: NCT04140331
Title: Level of Accelerometer-assessed Preoperative Physical Activity and Short Term Outcome After Elective Cardiac Surgery. A Monocentric Prospective Observational Cohort Study
Brief Title: Level of Accelerometer-assessed Preoperative Physical Activity and Short Term Outcome After Elective Cardiac Surgery
Acronym: ACTI-CARD
Status: Terminated | Type: Observational
Why Stopped: Recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 19CH049; 2019-A00525-52 (Other: ANSM)
Record Dates: First submitted 2019-10-24; First posted 2019-10-25 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Heart Diseases
Keywords: Post-operative evolution; Accelerometer; Cardiac surgery; Accelerometry; Preoperative physical activity
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- complicated post-operative evolution: Patients with a postoperative intensive care unity length of stay ≥ 5 days after elective cardiac surgery. They will have an accelerometer.
  Interventions: Device: Accelerometer
- simple post-operative evolution: Patients with a postoperative intensive care unity length of stay < 5 days after elective cardiac surgery. They will have an accelerometer.
  Interventions: Device: Accelerometer

INTERVENTIONS:
Device: Accelerometer — Patient will wear the accelerometer for 7 consecutive days to measure the level of physical activity.

SUMMARY:
Short term morbidity after elective cardiac surgery remains significant. Standard predictive models, considering simple patient demographics and clinical parameters, show limited efficiency in individual operative risk assessment. There is growing evidence about daily physical activity as a relevant indicator of preoperative "frailty". Although cardiopulmonary exercise testing remains a gold standard, we are looking for more simple tools in order to identify patients with poor physical condition. Accelerometry may be an objective and reproductible method to measure physical activity at patient's home.

DETAILED DESCRIPTION:
The aim of this study is to compare accelerometer-assessed preoperative physical activity between two groups of patients with different postoperative length of stay following elective cardiac surgery. In the future, accelerometry could be used to identify patients that may benefit from prehabilitation programs including exercise therapy before elective cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (≥ 60 years) awaiting elective cardiac surgery
* Patients affiliated or entitled to a social security scheme
* Patients who have received information about the study and have given their oral consent to participate

Exclusion Criteria:

* Pregnant woman,
* Major limitations in physical activity for orthopedic or musculoskeletal reasons
* Patients under judicial protection (curator or guardianship)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subject (≥ 60 years) awaiting elective cardiac surgery will be included.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Mean daily preoperative walking activity (average of steps/day over a period of 7 days) | Day: 7
  Measured by accelerometry.

SECONDARY OUTCOMES:
Total energy expenditure evaluated over a 7 days (steps/day) | Day: 7
  Measured by accelerometry.
Low activity time in hours per week (hours/week) | Day: 7
  Measured by accelerometry.
Moderate activity time in hours per week (hours/week) | Day: 7
  Measured by accelerometry.
Intense activity time in hours per week (hours/week) | Day: 7
  Measured by accelerometry.
Time of very intense activity in hours per week (hours/week) | Day: 7
  Measured by accelerometry.
Sleep time in hours per week (hours/week) | Day: 7
  Measured by accelerometry.
Analysis of questionary Duke Activity Status Index (DASI) over a period of 7 days | Day: 7
  Questionary Duke Activity Status Index (DASI) estimates the maximum volume of oxygen used in one minute (VO2 Max) as well as its effort capacity in metabolic equivalent.
  It contains 11 items. The higher the score indicates better functional capacity.
Analysis of questionary Short Nutritional Assessment Questionnaire (SNAQ) over a period of 7 days | Day: 7
  Questionary Short Nutritional Assessment Questionnaire (SNAQ) evaluates nutritional status. The higher the score indicates an important nutritional support.
Dosage of albumin (g/L) | Day: 7
  Measured by blood sample.
Dosage of prealbumin (g/L) | Day: 7
  Measured by blood sample.
Preoperative strength assessed by dynamometry (Kg) | Day: 14
  Measured by Hand Grip test.
Relationship between preoperative physical activity and duration of stay in intensive care | Months: 26
  Correlation between preoperative physical activity and duration of stay in intensive care.
Preoperative clinical outcome and duration of stay in intensive care | Months: 26
  Correlation between preoperative clinical outcome and duration of stay in intensive care.
Postoperative clinical outcome and duration of stay in intensive care | Months: 26
  Correlation between postoperative clinical outcome and duration of stay in intensive care.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles PALAO, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No